CLINICAL TRIAL: NCT02718144
Title: A Phase I/II Clinical Trial Assessing Safety and Efficacy of Estetrol (E4) in Postmenopausal Women With Advanced Estrogen Receptor Positive (ER+) Breast Cancer
Brief Title: Assessment of Safety and Efficacy of Estetrol in Postmenopausal Women With Advanced Estrogen Receptor Positive (ER+) Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pantarhei Oncology B.V. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR3106
Record Dates: First submitted 2016-03-02; First posted 2016-03-24 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2019-11

CONDITIONS: Breast Neoplasms
Keywords: dose-escalation; safety; dose-limiting toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- estetrol (Experimental): 3 + 3 design with inter-patient dose escalation
  Interventions: Drug: Estetrol

INTERVENTIONS:
Drug: Estetrol — Estetrol formulated in tablets, in escalating doses, will be investigated in patients with estrogen receptor positive (ER+) locally advanced or metastatic breast cancer.

SUMMARY:
This is a multi-center, open-label, phase I/IIa trial, dose-escalation study with a 3 + 3 cohort design to determine the recommended dose of estetrol for the treatment of patients with advanced breast cancer. After completing phase I part of the study (i.e. 4 weeks of treatment), patients will receive further treatment for 8 weeks at their individual phase I dose level (phase IIa part of the study).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with ER-positive and HER2-negative locally advanced and/or metastatic breast cancer, who progressed on standard therapies or for whom standard therapies are intolerant;
* Patients should have experienced a natural or surgical menopause at least 5 years ago;
* Failure of anti-estrogen treatment with tamoxifen and aromatase inhibitor(s) due to the development of resistance or unacceptable side effects with this treatment;
* No undiagnosed vaginal bleeding;
* No treatment with fulvestrant within 6 months of start of treatment;
* Life expectancy at least 6 months;
* Tumour assessment (CT scan) before the start of the E4 treatment;
* Body mass index (BMI) between (≥) 18 and (≤) 35 kg/m2;
* Able to swallow an oral medication;
* Acceptable values of hematological parameters, liver and kidney function and calcium levels;
* Acceptable values of hemostasis parameters (as of second cohort);
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-2 (as of second cohort);
* Reasonable physical and mental health as judged by the investigator and determined by physical examination, clinical laboratory assessments and vital signs;
* Willing to give informed consent in writing.

Exclusion Criteria:

* Uncontrolled nausea, vomiting, or diarrhea;
* History of venous or arterial thromboembolic disease or a known defect in the blood coagulation system;
* History of severe cardiac events or life threatening cardiac dysrhythmia (as of second cohort);
* Patients who have unstable angina or clinical congestive heart failure (as of second cohort);
* Uncontrolled hypertension, i.e. systolic blood pressure 160 mmHg and/or diastolic blood pressure 100 mmHg in the last 6 months with or without medication;
* Diabetes mellitus with poor glycaemic control in the last 6 months (HbA1c above 7.5%);
* Any other serious disease including systemic lupus erythematosus and untreated cholelithiasis;
* Smoking >10 cigarettes/day;
* Use of any other cancer therapy including radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy, chemotherapy, or use of other investigational agents at the start of treatment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The number of patients with a dose limiting toxicity (DLT) | 4 weeks

SECONDARY OUTCOMES:
Questionnaire on estrogen deficiency symptoms | 12 weeks
  Quality of Life will be assessed by means of a questionnaire on estrogen deficiency symptoms.
Pharmacokinetics: estetrol trough levels | 2 weeks, 4 weeks, 8 weeks
Preliminary anti-tumour response according to RECIST 1.1 | 12 weeks

OTHER OUTCOMES:
Number of patients with Adverse Events (AEs) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Katholisches Klinikum Mainz, Mainz
  - Universitatsmedizin Mainz, Mainz

REFERENCES:
- [Result] Singer CF, Bennink HJ, Natter C, Steurer S, Rudas M, Moinfar F, Appels N, Visser M, Kubista E. Antiestrogenic effects of the fetal estrogen estetrol in women with estrogen-receptor positive early breast cancer. Carcinogenesis. 2014 Nov;35(11):2447-51. doi: 10.1093/carcin/bgu144. Epub 2014 Jul 5. PMID 24997853
- [Result] Visser M, Kloosterboer HJ, Bennink HJ. Estetrol prevents and suppresses mammary tumors induced by DMBA in a rat model. Horm Mol Biol Clin Investig. 2012 Apr 1;9(1):95-103. doi: 10.1515/hmbci-2012-0015. PMID 25961355